CLINICAL TRIAL: NCT00940407
Title: A Pilot Study to Evaluate Clinical Outcomes of Photobiomodulation in Patients With Age Related Macular Degeneration of the Dry Type.
Brief Title: Toronto and Oak Ridge Photobiomodulation Study for Dry Age Related Macular Degeneration
Acronym: TORPA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merry, Graham, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOPRPA 08001
Record Dates: First submitted 2009-07-14; First posted 2009-07-16 (Estimated); Last update posted 2011-11-18 (Estimated); Status verified 2011-11

CONDITIONS: Nonexudative Age-related Macular Degeneration
Keywords: dry AMD; light treatment; ARMD; photobiomodulation; macular; eye disease; ageing eye disease
MeSH Terms: conditions — Eye Diseases | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Photobiomodulation (Gentlewaves, Warp 10) — Two separate light emitting devices that are already approved for other indications are used. Treatment will consist of 18 treatments lasting approximately two minutes per treatment.
  Other Names: Gentlewaves; Warp 10

SUMMARY:
The purpose of this study is to evaluate clinical outcomes of Photobiomodulation treatment on patients with dry Age Related Macular Degeneration (AMD).

Photobiomodulation is the use of non thermal, non laser light of specific wavelengths and energy directly on the eye to improve retinal function and delay AMD progression.

This is a prospective 2 center phase 2 clinical pilot study with no placebo group.

DETAILED DESCRIPTION:
Dry AMD is a progressive sight threatening disease affecting central acute vision. Dry AMD may progress to the wet form where leaking and bleeding in the retina can cause sudden severe visual loss.

There are no proven active treatments for Dry AMD. Dry AMD accounts for over 80% of AMD cases.

There are estimated to be 30 million people afflicted with AMD by the year 2020 in North America.

Photobiomodulation in this study is utilised by using two devices that are already approved for other indications by the FDA and Health Canada.

Photobiomodulation is a novel clinical application for treating dry AMD. As this is a pilot study there is no placebo or control group.

ELIGIBILITY:
Inclusion Criteria:

* patients of both genders aged 50 years inclusive and over
* patients must have DRY macular degeneration in the study eye
* best corrected visual acuity between 20/40 and 20/200
* patients must be competent to sign and have signed a consent form before study entry

Exclusion Criteria:

* visually significant cataracts
* presence of a visually significant posterior capsule if prior cataract has been performed
* any visually significant disease process in any ocular structure that would affect vision unrelated to macular degeneration
* a patient can be enrolled if only one of their eyes meets the criteria
* patients with severe clinically significant medical disease or unstable medical conditions including cardiovascular, hepatic, renal, neurological, endocrine, gastrointestinal, CNS or life threatening disease or current malignancy at the discretion of the investigators
* patients who are non-ambulatory or bed ridden
* female patients who are pregnant or of childbearing potential as the effects of PBM on the developing fetus are unknown
* patients with a history of epilepsy
* patients with a history of alcohol, drug or substance abuse in the past 6 months
* patients deemed uncooperative or non compliant with the requirements of the protocol
* patients who have received any investigational drug or treatment within 30 days prior to study entry
* patients who are not competent to understand and sign consent form

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Change in ETDRS Visual Acuity | prior to intervention and 3 monthly intervals to 1 year

SECONDARY OUTCOMES:
change in contrast sensitivity | prior to intervention and 3 monthly to 1 year
changes in retinal function parameters from Nidek MP1 assessment | prior to intervention and 3 monthly to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Graham F Merry, MBBS; LMCC, Principal Investigator — Dr. Graham Merry; Robert Dotson, M.D., Principal Investigator — Dr. Robert Dotson
Locations (2):
- Dr Robert Dotson, Oak Ridge, Tennessee, United States
- Dr Graham Merry, Toronto, Ontario, Canada